CLINICAL TRIAL: NCT02171715
Title: Relative Bioavailability of a Single Dose 20 mg BIBW 2992 Administered as Tablet (Final Formulation) Compared to BIBW 2992 Drinking Solution and BIBW 2992 Tablet (Trial Formulation II) Following Oral Administration to Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Three-way Crossover Phase I Study)
Brief Title: BIBW 2992 Administered as Tablet (Final Formulation) Compared to BIBW 2992 Drinking Solution and BIBW 2992 Tablet (Trial Formulation II) in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1200.35
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Afatinib

ARMS (3):
- BIBW 2992 MA2, final formulation (Experimental)
  Interventions: Drug: BIBW 2992 MA2
- BIBW 2992 MA2, trial formulation II (Experimental)
  Interventions: Drug: BIBW 2992 MA2
- BIBW 2992 MA 2 drinking solution (Active Comparator)
  Interventions: Drug: BIBW 2992 MA2

INTERVENTIONS:
Drug: BIBW 2992 MA2 — film-coated immediate release tablet - final formulation
  Arms: BIBW 2992 MA2, final formulation
Drug: BIBW 2992 MA2 — film-coated immediate release tablet - trial formulation II
  Arms: BIBW 2992 MA2, trial formulation II
Drug: BIBW 2992 MA2 — powder for oral solution
  Arms: BIBW 2992 MA 2 drinking solution

SUMMARY:
The primary objective of the study was to investigate the relative bioavailability and pharmacokinetics of 20 mg BIBW 2992 administered as film-coated immediate release tablet (final formulation, i.e. phase III/to-be-marketed formulation) to healthy subjects in comparison with the drinking solution and in comparison with the trial formulation II tablet, which was administered in phase II clinical trials and also partly in phase I trials.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to a complete medical history, including a physical examination, vital signs (BP (blood pressure), PR (pulse rate)), 12-lead ECG (electrocardiogram), and clinical laboratory tests
* Age 21 to 55 years, inclusive
* Body mass index 18.5 to 29.9 kg/m2, inclusive
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including drug allergy or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within one month prior to administration of the trial drug or during the trial
* Use of any drugs (including herbal preparations, vitamins and nutrient supplements) within 10 days prior to first administration of the trial drug or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking within the in-house periods from 12 hours before until 25 hours after each administration of the trial drug
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration of the trial drug or during the trial)
* Excessive physical activities (within one week prior to administration of the trial drug or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de Points, e.g., heart failure, hypokalemia, family history of Long QT Syndrome

Exclusion criteria specific for this study:

* Total bilirubin greater than 1.5 mg/dL
* History of clinically relevant skin diseases, psoriasis or moderate/severe acne
* Female gender
* Male subjects who refuse to minimise the risk of female partners becoming pregnant from the first dosing day until 3 months after the completion of the study. Acceptable methods of contraception for male volunteers include a vasectomy no less than 3 months prior to dosing, barrier contraception or another medically accepted contraceptive method. For female partners of male volunteers, acceptable methods of contraception include intrauterine device, tubal ligation, hormonal contraceptive for at least two months, or diaphragm with spermicide

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 96 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | up to 96 hours after drug administration

SECONDARY OUTCOMES:
AUC (area under the concentration-time curve of the analyte in plasma) for several time points | up to 96 hours after drug administration
%AUCtz-∞ (percentage of the AUCtz-∞ that is obtained by extrapolation from the last quantifiable data point to infinity) | up to 96 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 96 hours after drug administration
λz (terminal rate constant in plasma) | up to 96 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | up to 96 hours after drug administration
MRTpo (mean residence time of the analyte in the body after oral administration) | up to 96 hours after drug administration
CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 96 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 96 hours after drug administration
Number of patients with adverse events | up to 88 days
Assessment of tolerability by the investigator on a 4-point scale | Day 5 of each treatment period